CLINICAL TRIAL: NCT04525131
Title: A Window of Opportunity Study to Characterize the Safety, Dose Tolerance, Pharmacokinetics, and Pharmacodynamics of CPX-POM in Patients With Newly Diagnosed or Recurrent Bladder Tumors
Brief Title: Safety, Dose Tolerance, Pharmacokinetics, Pharmacodynamics of CPX-POM in Patients With Newly Diagnosed or Recurrent Bladder Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CicloMed LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPX-POM-002
Record Dates: First submitted 2020-08-11; First posted 2020-08-25 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Bladder Cancer
Keywords: Newly diagnosed or recurrent bladder tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPX-POM (Experimental): IV over 20 minutes once per day
  Interventions: Drug: CPX-POM

INTERVENTIONS:
Drug: CPX-POM — CPX-POM

SUMMARY:
This is a phase II, single center open label to determine safety, dose tolerance, PK and PD of the recommended Phase 2 dose (RP2D) of CPX-POM administered in patients with any newly diagnosed or recurrent bladder tumors.

DETAILED DESCRIPTION:
This will be an open-label study to determine the safety, dose tolerance, pharmacokinetics, and pharmacodynamics of CPX-POM in patients with newly diagnosed or recurrent, untreated or intravesical treatment completed >6 months before the current diagnosis, resectable tumors. Approximately 12 patients will be enrolled and treated with 900 mg/m2 CPX-POM administered IV over 20 minutes once per day for 5 days followed by TURBT on Day 5 after the fifth dose. TURBT will be performed 2 to 6 hours following drug administration on Day 5.

Pretreatment bladder tumor tissues will be obtained at the time of in-office cystoscopy by cold cup biopsy within 4 weeks of TURBT. Posttreatment bladder tumor tissues will be obtained at TURBT. Bladder tumor tissues will undergo pathological evaluation at each site.

Prior to administration of the first CPX-POM dose on Day 1, pre-dose blood (plasma) and urine (clean catch) samples will be collected. At the time of TURBT on Day 5, one 3-mL blood (plasma) sample and a urine specimen will be collected for measurement of CPX-POM concentrations.

Patients will be followed for at least 30 days after the last dose of CPX-POM for safety

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female aged ≥18 years.
2. Patient provided signed and dated informed consent prior to initiation of any study procedures.
3. Patient is likely to have a new bladder tumor based on clinical presentation or is at high risk for tumor recurrence based on previous history.
4. Patient has a cystoscopically confirmed bladder tumor and will be scheduled to undergo TURBT.
5. Patient has not received prior treatment for bladder cancer or completed their last intravesical therapy >6 months before screening.
6. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 (fully active, able to carry out all pre-disease activities without restriction) or 1 (unable to perform physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
7. Patient has a predicted life expectancy of ≥3 months.
8. Patient has adequate renal function (creatinine ≤1.5 × the upper limit of the normal range (ULN) or an estimated glomerular filtration rate (eGFR) of >30 mL/min/1.73 m2).
9. Patient has adequate hepatic function, as evidenced by a total bilirubin ≤1.5 × ULN, aspartate aminotransferase (AST) ≤3 × ULN and /or alanine aminotransferase (ALT) ≤3 × ULN.
10. Patient has adequate bone marrow function, as evidenced by hemoglobin ≥9.0 g/dL in the absence of transfusion within the previous 72 hours, platelet count ≥100×10^9cells/L, and absolute neutrophil count (ANC) ≥1.5×10^9 cells/L.
11. Patient has no significant ischemic heart disease or myocardial infarction within 6 months before the first dose of CPX-POM and currently has adequate cardiac function, as evidenced by a left ventricular ejection fraction of >50% as assessed by multi-gated acquisition (MUGA) or ultrasound/echocardiography (ECHO); and corrected QT interval by Fridericia's correction formula (QTcF) <450 msec for males and <470 msec for females. The eligibility of patients with ventricular pacemakers for whom the QT interval may not be accurately measurable will be determined on a case-by-case basis by the Sponsor in consultation with the Medical Monitor.
12. Patient and his/her partner agree to use adequate contraception after providing written informed consent through 3 months after the last dose of CPX-POM, as follows:

    1. For women: Negative pregnancy test during Screening and at Day 1 of each treatment cycle and compliant with a medically-approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile or postmenopausal.
    2. For men: Compliant with a medically-approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile. Men whose sexual partners are of child-bearing potential must agree to use 2 methods of contraception prior to study entry, during the study, and for 3 months after the treatment period.
13. Patient is willing and able to participate in the study and comply with all study requirements.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Patients received prior intravesical therapy for bladder cancer within ≤6 months of the current diagnosis.
2. Patients must not have had any of the following within 6 months before study drug administration:

   1. Myocardial infarction
   2. Severe/unstable angina
   3. Symptomatic congestive heart failure
   4. Cerebrovascular accident or transient ischemic attack, or
   5. Pulmonary embolism
3. Ongoing cardiac dysrhythmias of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 grade 2.
4. Evidence of New York Heart Association (NYHA) functional class III or IV heart disease.
5. Uncontrolled hypertension (>150/100 mmHg despite optimal medical therapy).
6. Patient has an uncontrolled or severe intercurrent medical condition. The decision to exclude a patient from the study for an uncontrolled or severe intercurrent medical condition will be made by the Principal Investigator. Examples could include epilepsy, resistant infection, or any other neurological disease that would make clinical assessment difficult.
7. Patient underwent major surgery or radiation therapy within 4 weeks before the first dose of CPX-POM or received an investigational drug or device within 4 weeks or 5 half-lives of that agent (whichever is shorter) before the first dose of CPX-POM. A minimum of 10 days between termination of the investigational drug and administration of CPX-POM is required.
8. If female, patient is pregnant or breast-feeding.
9. Patient has evidence of a serious active infection (e.g., infection requiring treatment with IV antibiotics).
10. Patient has a known, active Hepatitis A infection.
11. Patient has known human immunodeficiency virus (HIV) or Hepatitis B, or C infection, as such patients may be at increased risk for toxicity due to concomitant treatment and disease-related symptoms may preclude accurate assessment of the safety of CPX POM.
12. Patient has an important medical illness or abnormal laboratory finding that, in the Investigator's opinion, would increase the risk of participating in this study.
13. Patient is taking warfarin.
14. Patients may not have another malignancy that could interfere with the evaluation of safety or efficacy of the study drug. Patients with a prior malignancy will be allowed without approval in the following circumstances:

    1. Not currently active and diagnosed at least 3 years prior to the date of registration.
    2. Non-invasive diseases such as low risk cervical cancer or any cancer in situ.
    3. Localized (early stage) cancer treated with curative intent (without evidence of recurrence and intent for further therapy), and in which no chemotherapy was indicated.(e.g., low/intermediate risk prostate cancer, etc.).
    4. Non-muscle invasive bladder cancer (NMIBC) for which treatment was completed >6 months before the current diagnosis.
15. Patient has known allergy or hypersensitivity to any component of CPX-POM.
16. Patient is taking any iron replacement therapy administered IV, intramuscularly, or orally due to the potential for loss of anticancer activity due to drug and/or metabolites chelating iron.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Taylor III, MD, MSc, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weir SJ, Dandawate P, Standing D, Bhattacharyya S, Ramamoorthy P, Rangarajan P, Wood R, Brinker AE, Woolbright BL, Tanol M, Ham T, McCulloch W, Dalton M, Reed GA, Baltezor MJ, Jensen RA, Taylor JA 3rd, Anant S. Fosciclopirox suppresses growth of high-grade urothelial cancer by targeting the gamma-secretase complex. Cell Death Dis. 2021 May 31;12(6):562. doi: 10.1038/s41419-021-03836-z. PMID 34059639

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CPX-POM
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | CPX-POM
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.41 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Serious Adverse Events (SAEs)
Description: Incidence of Serious Adverse Events in subjects receiving CPX-POM as assessed by (CTCAE) version 5.0
Time Frame: 35 days
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-POM
Number analyzed (Participants) | 12
Participants | 1

2. Primary Outcome: Number of Participants With Any Adverse Events (AEs)
Description: Incidence of Adverse Events in subjects receiving CPX-POM as assessed by (CTCAE) version 5.0
Time Frame: 35 days
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-POM
Number analyzed (Participants) | 12
Participants | 9

3. Primary Outcome: Evaluate the Dose Limiting Toxicities (DLTs) of CPX-POM
Description: A DLT will include some Grade 3 or 4 AEs if deemed related to study drug. In addition, any patient who is unable to receive 80% of the expected dose of CPX-POM (i.e., patients who are unable to receive at least 4 of the 5 scheduled doses) because of AEs will be considered to have a DLT.
Time Frame: 35 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-POM
Number analyzed (Participants) | 12
Participants | 2

4. Secondary Outcome: Incidence of Treatment Related Adverse Events
Description: To determine the number of subjects with treatment related AEs
Time Frame: 35 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-POM
Number analyzed (Participants) | 12
Participants | 4

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | CPX-POM
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPX-POM (N=12)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPX-POM (N=12)
Dizziness (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Fatigue (General disorders) | 2
Gait disturbance (General disorders) | 1
Injection site reaction (General disorders) | 1
Confusional state (Psychiatric disorders) | 3
Hypertension (Vascular disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor and the PI plan to publish the data.

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT04525131/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT04525131/SAP_001.pdf